CLINICAL TRIAL: NCT06354413
Title: Establishing a Database of Patients Undergoing Surgery for Hypertrophic Cardiomyopathy (Concomitant Bypass Surgery)
Brief Title: Outcomes of Concomitant Bypass Surgery in Septal Myectomy
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Shuiyun Wang, Dr., Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2023-2261
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Hypertrophic Cardiomyopathy; Coronary Artery Disease; Myocardial Bridging
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Coronary Artery Disease; Myocardial Bridging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CABG during myectomy — To explore the effect of CABG during myectomy. No control group

SUMMARY:
To investigate clinical characteristics and survival outcomes of patients with obstructive hypertrophic cardiomyopathy who underwent concomitant coronary artery bypass grafting during septal myectomy.

DETAILED DESCRIPTION:
Surgical septal myectomy (SM) is an effective approach for treating patients with drug-refractory obstructive hypertrophic cardiomyopathy (HCM).However, numerous patients with HCM exhibit concurrent ischemic heart disease, including atherosclerotic coronary artery disease (CAD) and myocardial bridging (MB). Although patients with HCM have been known to possess diminished coronary flow reserve,additional CAD can worsen myocardial ischemia, contributing to an unfavorable prognosis.MB, although infrequent, may affect diastolic heart perfusion, leading to angina and even sudden death.Current guidelines recommend revascularization for ischemic heart disease caused by CAD and MB.However, the impact of concomitant coronary revascularization during HCM management remains unclear. In this study, we analyzed the clinical characteristics and surgical scenarios of patients who underwent concomitant coronary artery bypass grafting (CABG) during ventricular SM and investigated their prognosis.

Patient clinical and survival data from 2009-2020 were retrospectively reviewed. The median follow-up period was 5.1 years. All-cause mortality was the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of obstructive hypertrophic cardiomyopathy.
2. Undergo ventricular septal resection and cardiac bypass surgery at the same time.

Exclusion Criteria:

Incomplete surgical and follow-up data

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with obstructive hypertrophic cardiomyopathy who underwent concomitant coronary artery bypass grafting(due to atherosclerosis coronary artery diseases or myocardial bridge) during septal myectomy.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | through study completion, an average of 5 year
  death because of any reason

SECONDARY OUTCOMES:
cardiac-related deaths and readmission | through study completion, an average of 5 year
  deaths and readmission because of heart failure, stoke, and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Lu, MD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: No